CLINICAL TRIAL: NCT00051038
Title: A Phase II Study of the Safety and Efficacy of Adding Entecavir to Current Lamivudine Therapy in HIV and HBV Co-Infected Patients Who Have Hepatitis B Viremia While Being Treated With Lamivudine
Brief Title: Study of Adding Entecavir to Current Lamivudine Therapy in HIV and HBV Co-Infected Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: AI463-038
Record Dates: First submitted 2002-12-31; First posted 2003-01-03 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2007-08

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — entecavir

INTERVENTIONS:
Drug: Entecavir

SUMMARY:
The purpose of this clinical research study is to assess the safety and effectiveness of entecavir, when being added to lamivudine, in the treatment of adults with chronic hepatitis B infection who are co-infected with HIV.

ELIGIBILITY:
* Documented history of co-infection with HIV and HBV
* Stable Anti Retroviral Therapy regimen containing lamivudine 150 mg BID for at least 24 weeks prior to enrollment;
* Documented HBV viremia on screening and at least at 4 weeks prior to screening
* HBe Ag-positive or HBe Ag-negative / anti-HBe-positive
* HIV viral load below 400 copies/mL by the Roche Amplicor(TM) 1.5 HIV PCR assay at screening and equally low at least 12 weeks prior to screening
* Absence of Co-Infection with hepatitis C virus (HCV) or hepatitis D virus (HDV)
* Absence of other forms of liver disease e.g., alcoholic, autoimmune, biliary disease
* Less that 1/2 weeks of prior therapy with nucleoside/nucleotide analogue (excluding lamivudine) with activity against HBV (including e.g. famciclovir, tenofovir, ganciclovir, adefovir). No receipt of any of these therapies within 24 weeks prior to randomization into this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Local Institution, New Haven, Connecticut
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Lousiville, Kentucky
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Pittsburgh, Pennsylvania